CLINICAL TRIAL: NCT00874432
Title: Effect of ACE-inhibitors on Aortic Stiffness in Elderly Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-2008-0221; A534280 (Other: UW Madison); SMPH/MEDICINE/NEPHROLOGY (Other: UW Madison)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Disease; Chronic Kidney Disease
Keywords: cardiovascular disease; angiotensin converting enzyme inhibitors; chronic kidney disease; cardiovascular disease in elderly patients with CKD
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic | interventions — Angiotensin-Converting Enzyme Inhibitors; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Chronic Kidney Disease-ACE-I (Active Comparator): ace inhibitor
  Interventions: Drug: lisinopril
- Chronic Kidney Disease (Placebo Comparator)
  Interventions: Drug: angiotensin converting enzyme inhibitor
- Age matched control-ACE-I (Active Comparator): ace-inhibitor
  Interventions: Drug: lisinopril
- Age matched control (Placebo Comparator): Placebo
  Interventions: Drug: angiotensin converting enzyme inhibitor

INTERVENTIONS:
Drug: angiotensin converting enzyme inhibitor — Active comparator in chronic kidney disease and age matched control will take 1x40mg per day Placebo comparator in chronic kidney disease and age matched control will take 1 placebo pill per day
  Other Names: ACE-inhibitor
  Arms: Age matched control; Chronic Kidney Disease
Drug: lisinopril — 1 x 40 mg per day
  Other Names: ace inhibitor
  Arms: Age matched control-ACE-I; Chronic Kidney Disease-ACE-I

SUMMARY:
The goal of this proposal is to investigate the potential for ACE-inhibitors (ACE-I)(drugs primarily used to treat hypertension or congestive heart failure) to prevent or delay cardiovascular disease (CVD) in older adults with chronic kidney disease (CKD) by examining their impact on aortic stiffness in people with stage 3 CKD in a randomized, controlled study.

DETAILED DESCRIPTION:
This study will be the first to examine whether aortic stiffness is increased in elderly patients with CKD compared to their age-matched healthy controls and further examine whether ACE-I may delay the progression of aortic stiffness in elderly CKD patients. If ACE-I therapy appears beneficial in preventing or delaying arterial stiffening in elderly patients with CKD, this work has important implications for improving the overall health of this population.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* BP 120/80 or higher *(bps will be checked weekly first 4 weeks to ensure < 130/80 - IF bp remains > 130/80 we will administer other bp meds per JNC VII guidelines)
* CKD stage 3 (GFR 30 - 59 ml/min) for CKD group; no CKD for control group

Exclusion Criteria:

* Known significant CVD (history of Myocardial infarction (MI), recurrent stroke, or New York Heart Association (NYHA) class III or greater).
* Serum potassium > 5.2 meq/L
* Known allergy or hypersensitivity to ACE inhibitor or ARB
* Female of childbearing age not practicing contraception
* Current treatment with an Angiotensin Converting Enzyme Inhibitors (ACE-I) or Angiotensin-Receptor Blockers (ARB) (Note: can participate if on ACE-I after 6 week washout period)
* History of ACE-I induced angioedema
* History of angioedema, hereditary or idiopathic
* Persons lacking consent capacity

  * 500 mg/dL proteinuria on 2 consecutive spot urine protein/creat ratios

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arjang Djamali, MD, Principal Investigator — University of Wisconsin-Madison School of Medicine and Public Health; Laura Maursetter, DO, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison Hospitals and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Ryan TP, Sloand JA, Winters PC, Corsetti JP, Fisher SG. Chronic kidney disease prevalence and rate of diagnosis. Am J Med. 2007 Nov;120(11):981-6. doi: 10.1016/j.amjmed.2007.05.012. PMID 17976426
- [Background] Foley RN, Parfrey PS. Cardiovascular disease and mortality in ESRD. J Nephrol. 1998 Sep-Oct;11(5):239-45. PMID 9831236
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, London GM. Arterial calcifications, arterial stiffness, and cardiovascular risk in end-stage renal disease. Hypertension. 2001 Oct;38(4):938-42. doi: 10.1161/hy1001.096358. PMID 11641313
- [Background] Covic A, Haydar AA, Bhamra-Ariza P, Gusbeth-Tatomir P, Goldsmith DJ. Aortic pulse wave velocity and arterial wave reflections predict the extent and severity of coronary artery disease in chronic kidney disease patients. J Nephrol. 2005 Jul-Aug;18(4):388-96. PMID 16245242
- [Background] London GM, Marchais SJ, Guerin AP. Arterial stiffness and function in end-stage renal disease. Adv Chronic Kidney Dis. 2004 Apr;11(2):202-9. doi: 10.1053/j.arrt.2004.02.008. PMID 15216492
- [Background] Wang MC, Tsai WC, Chen JY, Huang JJ. Stepwise increase in arterial stiffness corresponding with the stages of chronic kidney disease. Am J Kidney Dis. 2005 Mar;45(3):494-501. doi: 10.1053/j.ajkd.2004.11.011. PMID 15754271
- [Background] Kundhal K, Lok CE. Clinical epidemiology of cardiovascular disease in chronic kidney disease. Nephron Clin Pract. 2005;101(2):c47-52. doi: 10.1159/000086221. Epub 2005 Jun 7. PMID 15942250
- [Background] Willum-Hansen T, Staessen JA, Torp-Pedersen C, Rasmussen S, Thijs L, Ibsen H, Jeppesen J. Prognostic value of aortic pulse wave velocity as index of arterial stiffness in the general population. Circulation. 2006 Feb 7;113(5):664-70. doi: 10.1161/CIRCULATIONAHA.105.579342. PMID 16461839
- [Background] London GM, Guerin AP, Marchais SJ, Pannier B, Safar ME, Day M, Metivier F. Cardiac and arterial interactions in end-stage renal disease. Kidney Int. 1996 Aug;50(2):600-8. doi: 10.1038/ki.1996.355. PMID 8840292
- [Background] Shinohara K, Shoji T, Tsujimoto Y, Kimoto E, Tahara H, Koyama H, Emoto M, Ishimura E, Miki T, Tabata T, Nishizawa Y. Arterial stiffness in predialysis patients with uremia. Kidney Int. 2004 Mar;65(3):936-43. doi: 10.1111/j.1523-1755.2004.00468.x. PMID 14871413
- [Background] Safar ME, London GM, Plante GE. Arterial stiffness and kidney function. Hypertension. 2004 Feb;43(2):163-8. doi: 10.1161/01.HYP.0000114571.75762.b0. Epub 2004 Jan 19. PMID 14732732
- [Background] Dao HH, Essalihi R, Bouvet C, Moreau P. Evolution and modulation of age-related medial elastocalcinosis: impact on large artery stiffness and isolated systolic hypertension. Cardiovasc Res. 2005 May 1;66(2):307-17. doi: 10.1016/j.cardiores.2005.01.012. PMID 15820199
- [Background] Ferrari AU, Radaelli A, Centola M. Invited review: aging and the cardiovascular system. J Appl Physiol (1985). 2003 Dec;95(6):2591-7. doi: 10.1152/japplphysiol.00601.2003. PMID 14600164
- [Background] Mitchell GF, Parise H, Benjamin EJ, Larson MG, Keyes MJ, Vita JA, Vasan RS, Levy D. Changes in arterial stiffness and wave reflection with advancing age in healthy men and women: the Framingham Heart Study. Hypertension. 2004 Jun;43(6):1239-45. doi: 10.1161/01.HYP.0000128420.01881.aa. Epub 2004 May 3. PMID 15123572
- [Background] Sawabe M, Takahashi R, Matsushita S, Ozawa T, Arai T, Hamamatsu A, Nakahara K, Chida K, Yamanouchi H, Murayama S, Tanaka N. Aortic pulse wave velocity and the degree of atherosclerosis in the elderly: a pathological study based on 304 autopsy cases. Atherosclerosis. 2005 Apr;179(2):345-51. doi: 10.1016/j.atherosclerosis.2004.09.023. Epub 2004 Dec 13. PMID 15777552
- [Background] London GM, Marchais SJ, Guerin AP, Pannier B. Arterial stiffness: pathophysiology and clinical impact. Clin Exp Hypertens. 2004 Oct-Nov;26(7-8):689-99. doi: 10.1081/ceh-200031982. PMID 15702623
- [Background] London GM, Marchais SJ, Guerin AP, Metivier F. Arteriosclerosis, vascular calcifications and cardiovascular disease in uremia. Curr Opin Nephrol Hypertens. 2005 Nov;14(6):525-31. doi: 10.1097/01.mnh.0000168336.67499.c0. PMID 16205470
- [Background] Touyz RM. The role of angiotensin II in regulating vascular structural and functional changes in hypertension. Curr Hypertens Rep. 2003 Apr;5(2):155-64. doi: 10.1007/s11906-003-0073-2. PMID 12642016
- [Background] Unger T. Pharmacological properties of angiotensin II antagonists: examining all the therapeutic implications. J Renin Angiotensin Aldosterone Syst. 2001 Sep;2 Suppl 2:S4-7. doi: 10.3317/jraas.2001.030. PMID 11881101
- [Background] Matsuda H, Hayashi K, Saruta T. Distinct time courses of renal protective action of angiotensin receptor antagonists and ACE inhibitors in chronic renal disease. J Hum Hypertens. 2003 Apr;17(4):271-6. doi: 10.1038/sj.jhh.1001543. PMID 12692572
- [Background] Chrysant SG. Vascular remodeling: the role of angiotensin-converting enzyme inhibitors. Am Heart J. 1998 Feb;135(2 Pt 2):S21-30. doi: 10.1053/hj.1998.v135.86971. PMID 9488609
- [Background] Bertrand ME. Provision of cardiovascular protection by ACE inhibitors: a review of recent trials. Curr Med Res Opin. 2004 Oct;20(10):1559-69. doi: 10.1185/030079904X4185. PMID 15462689
- [Background] Fields LE, Burt VL, Cutler JA, Hughes J, Roccella EJ, Sorlie P. The burden of adult hypertension in the United States 1999 to 2000: a rising tide. Hypertension. 2004 Oct;44(4):398-404. doi: 10.1161/01.HYP.0000142248.54761.56. Epub 2004 Aug 23. PMID 15326093
- [Background] Vasan RS, Beiser A, Seshadri S, Larson MG, Kannel WB, D'Agostino RB, Levy D. Residual lifetime risk for developing hypertension in middle-aged women and men: The Framingham Heart Study. JAMA. 2002 Feb 27;287(8):1003-10. doi: 10.1001/jama.287.8.1003. PMID 11866648
- [Background] Franklin SS, Gustin W 4th, Wong ND, Larson MG, Weber MA, Kannel WB, Levy D. Hemodynamic patterns of age-related changes in blood pressure. The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):308-15. doi: 10.1161/01.cir.96.1.308. PMID 9236450
- [Background] Lloyd-Jones DM, Evans JC, Levy D. Hypertension in adults across the age spectrum: current outcomes and control in the community. JAMA. 2005 Jul 27;294(4):466-72. doi: 10.1001/jama.294.4.466. PMID 16046653
- [Background] Hansson L, Zanchetti A, Carruthers SG, Dahlof B, Elmfeldt D, Julius S, Menard J, Rahn KH, Wedel H, Westerling S. Effects of intensive blood-pressure lowering and low-dose aspirin in patients with hypertension: principal results of the Hypertension Optimal Treatment (HOT) randomised trial. HOT Study Group. Lancet. 1998 Jun 13;351(9118):1755-62. doi: 10.1016/s0140-6736(98)04311-6. PMID 9635947
- [Background] Darne B, Girerd X, Safar M, Cambien F, Guize L. Pulsatile versus steady component of blood pressure: a cross-sectional analysis and a prospective analysis on cardiovascular mortality. Hypertension. 1989 Apr;13(4):392-400. doi: 10.1161/01.hyp.13.4.392. PMID 2522417
- [Background] Mitchell GF, Lacourciere Y, Ouellet JP, Izzo JL Jr, Neutel J, Kerwin LJ, Block AJ, Pfeffer MA. Determinants of elevated pulse pressure in middle-aged and older subjects with uncomplicated systolic hypertension: the role of proximal aortic diameter and the aortic pressure-flow relationship. Circulation. 2003 Sep 30;108(13):1592-8. doi: 10.1161/01.CIR.0000093435.04334.1F. Epub 2003 Sep 15. PMID 12975261
- [Background] Hallan S, Asberg A, Lindberg M, Johnsen H. Validation of the Modification of Diet in Renal Disease formula for estimating GFR with special emphasis on calibration of the serum creatinine assay. Am J Kidney Dis. 2004 Jul;44(1):84-93. doi: 10.1053/j.ajkd.2004.03.027. PMID 15211442
- [Background] Levey AS, Eckardt KU, Tsukamoto Y, Levin A, Coresh J, Rossert J, De Zeeuw D, Hostetter TH, Lameire N, Eknoyan G. Definition and classification of chronic kidney disease: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2005 Jun;67(6):2089-100. doi: 10.1111/j.1523-1755.2005.00365.x. PMID 15882252
- [Background] McEniery CM, Yasmin, Hall IR, Qasem A, Wilkinson IB, Cockcroft JR; ACCT Investigators. Normal vascular aging: differential effects on wave reflection and aortic pulse wave velocity: the Anglo-Cardiff Collaborative Trial (ACCT). J Am Coll Cardiol. 2005 Nov 1;46(9):1753-60. doi: 10.1016/j.jacc.2005.07.037. Epub 2005 Oct 10. PMID 16256881
- [Background] Mitchell GF, Izzo JL Jr, Lacourciere Y, Ouellet JP, Neutel J, Qian C, Kerwin LJ, Block AJ, Pfeffer MA. Omapatrilat reduces pulse pressure and proximal aortic stiffness in patients with systolic hypertension: results of the conduit hemodynamics of omapatrilat international research study. Circulation. 2002 Jun 25;105(25):2955-61. doi: 10.1161/01.cir.0000020500.77568.3c. PMID 12081987
- [Background] Bakris GL, Weir MR. Angiotensin-converting enzyme inhibitor-associated elevations in serum creatinine: is this a cause for concern? Arch Intern Med. 2000 Mar 13;160(5):685-93. doi: 10.1001/archinte.160.5.685. PMID 10724055
- [Background] Djamali A, Sadowski E, Muehrer R, et al. Losartan Improves Renal Medullary Oxygenation and Oxidative Stress in Patients with Chronic Allograft Nephropathy. J.Am.Soc.Nephrol. 15 (Abstract Issue):SA-PO1026, 2004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between January 2009 and May 2009. Patients were told about this study from the nephrologist or study coordinator around the time of their usual kidney clinic visit. Controls were enrolled through a group on campus who connects volunteers with research studies.
Pre-assignment Details: There is limited data for this study, the PI is now in private practice and some raw data no longer exists to answer this outcome. We have done our due diligence to populate this record with data that remains.
Period: Overall Study
Arm/Group | Chronic Kidney Disease-ACE-I | Chronic Kidney Disease | Age Matched Control-ACE-I | Age Matched Control
Started | 8 | 4 | 17 | 14
Completed | 5 | 2 | 9 | 11
Not Completed | 3 | 2 | 8 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Other | 1 | 2 | 8 | 3

BASELINE CHARACTERISTICS:
Population: Only data for Aim 1 of this study has been located.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease-ACE-I | Chronic Kidney Disease | Age Matched Control-ACE-I | Age Matched Control | Total
Number analyzed (Participants) | 8 | 4 | 17 | 14 | 43
Age, Continuous [Mean (Full Range); unit: years] | 65 [63 to 68] | 87 [74 to 90] | 63.4 [61 to 75] | 67.3 [62 to 79] | 68 [61 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 13 | 11 | 28
  Male | 5 | 3 | 4 | 3 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8 | 4 | 17 | 14 | 43
Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.3 (0.3) | 0.8 (1.8) | NA (NA) — data no longer exists | NA (NA) — data no longer exists | NA (NA) — unable to calculate

OUTCOME MEASURES:

1. Primary Outcome: Aortic Pulse Wave Velocity (PWV)
Description: PWV will be measured in patients over age 60 with stage 3 CKD and age matched controls without CKD.
Time Frame: up to 12 months
Population: Comparison of the baseline pulse wave velocity measures between the two groups (CKD vs no CKD) prior to intervention with ACE inhibitor. Data analyzed is from 32 participants due to drop out either from study self withdrawal (3) or ineligibility (1 = BP too low to start medication) and 7 without adequate testing data available for analysis.
Measure: Mean (Standard Deviation); unit: m/s
Groups:
- Chronic Kidney Disease: Participants over age 60 with Chronic Kidney Disease (CKD)
- Age Matched Control: Healthy age-matched control over age 60
Arm/Group | Chronic Kidney Disease | Age Matched Control
Number analyzed (Participants) | 11 | 22
m/s
  Carotid-Femoral Pulse Wave Velocity | 9.90 (1.12) | 9.96 (2.52)
  Carotid-Brachial Pulse Wave Velocity: number analyzed (Participants) | 11 | 21
  Carotid-Brachial Pulse Wave Velocity | 7.62 (1.76) | 8.57 (1.46)
  Carotid-Radial Pulse Wave Velocity | 9.03 (2.12) | 8.38 (1.76)
Statistical Analysis 1: Comparison: Chronic Kidney Disease vs Age Matched Control; p-value for CBPWV between CKD and Control groups; Test type: Superiority; p = 0.685, t-test, 2 sided
Statistical Analysis 2: Comparison: Chronic Kidney Disease vs Age Matched Control; p-value for CRPWV between CKD and Control groups; Test type: Superiority; p = 0.739, t-test, 2 sided
Statistical Analysis 3: Comparison: Chronic Kidney Disease vs Age Matched Control; p-value for CFPWV between CKD and Control groups; Test type: Superiority; p = 0.471, t-test, 2 sided

2. Secondary Outcome: Mean Vascular Stiffness As Measured by PWV
Description: Comparison between Participants with Stage 3 Chronic Kidney Disease (CKD) and age matched Controls without CKD. The numbers reported are the mean of all the participants in the group at two points in time - the baseline and at 12 months for CFPWV, CBPWV, and CRPWV.
  Carotid-Femoral Pulse Wave Velocity (CFPWV) Carotid-Brachial Pulse Wave Velocity (CBPWV) Carotid-Radial Pulse Wave Velocity (CRPWV)
Time Frame: baseline and 12 months
Population: Participants in each arm that had measurements for both baseline and 12 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Chronic Kidney Disease-ACE-I | Chronic Kidney Disease | Age Matched Control-ACE-I | Age Matched Control
Number analyzed (Participants) | 5 | 1 | 10 | 11
m/s
  CBPWV Baseline | 7.87 (1.70) | 6.28 (NA) — only one measurement | 9.14 (0.82) | 8.17 (1.61)
  CBPWV 12 months | 8.40 (2.50) | 8.28 (0.54) | 8.65 (1.87) | 8.06 (2.02)
  CRPWV Baseline | 9.03 (0.93) | 4.80 (NA) — only one measurement | 9.75 (0.95) | 8.95 (1.69)
  CRPWV 12 months | 8.57 (2.03) | 8.66 (2.87) | 8.16 (1.93) | 9.43 (1.71)
  CFPWV Baseline | 10.20 (0.99) | 7.95 (NA) — only one measurement | 9.96 (2.52) | 9.55 (2.64)
  CFPWV 12 months | 11.07 (2.29) | 10.66 (2.78) | 8.33 (1.06) | 9.79 (1.97)
Statistical Analysis 1: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the baseline CBPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.685, t-test, 2 sided
Statistical Analysis 2: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the 12 month CBPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.869, t-test, 2 sided
Statistical Analysis 3: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the baseline CRPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.709, t-test, 2 sided
Statistical Analysis 4: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the 12 month CBPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.340, t-test, 2 sided
Statistical Analysis 5: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the baseline CFPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.730, t-test, 2 sided
Statistical Analysis 6: Comparison: Chronic Kidney Disease vs Age Matched Control; This p-value compares the 12 month CFPWV measures for the CKD vs Controls group; Test type: Superiority; p = 0.204, t-test, 2 sided
Statistical Analysis 7: Comparison: Chronic Kidney Disease-ACE-I vs Age Matched Control-ACE-I; This compares the 12 month CBPWV measure of ACE-I CKD and Control groups; Test type: Superiority; p = 0.963, t-test, 2 sided
Statistical Analysis 8: Comparison: Chronic Kidney Disease-ACE-I vs Age Matched Control-ACE-I; This compares the 12 month CRPWV measure of ACE-I CKD and Control groups; Test type: Superiority; p = 0.991, t-test, 2 sided
Statistical Analysis 9: Comparison: Chronic Kidney Disease-ACE-I vs Age Matched Control-ACE-I; This compares the 12 month CFPWV measure of ACE-I CKD and Control groups; Test type: Superiority; p = 0.176, t-test, 2 sided
Statistical Analysis 10: Comparison: Chronic Kidney Disease-ACE-I; This compares the baseline and 12 month CBPWV measure of the ACE-I CKD; Test type: Superiority; p = 0.402, t-test, 2 sided
Statistical Analysis 11: Comparison: Chronic Kidney Disease-ACE-I; This compares the baseline and 12 month CRPWV measure of the ACE-I CKD; Test type: Superiority; p = 0.586, t-test, 2 sided
Statistical Analysis 12: Comparison: Chronic Kidney Disease-ACE-I; This compares the baseline and 12 month CFPWV measure of the ACE-I CKD; Test type: Superiority; p = 0.455, t-test, 2 sided
Statistical Analysis 13: Comparison: Age Matched Control-ACE-I; This compares the baseline and 12 month CBPWV measure of the ACE-I Control Group; Test type: Superiority; p = 0.418, t-test, 2 sided
Statistical Analysis 14: Comparison: Age Matched Control-ACE-I; This compares the baseline and 12 month CRPWV measure of the ACE-I Control Group; Test type: Superiority; p = 0.091, t-test, 2 sided
Statistical Analysis 15: Comparison: Age Matched Control-ACE-I; This compares the baseline and 12 month CFPWV measure of the ACE-I Control Group; Test type: Superiority; p = 0.034, t-test, 2 sided
Statistical Analysis 16: Comparison: Chronic Kidney Disease vs Age Matched Control; This compares the 12 month CBPWV measure of the CKD and Control groups; Test type: Superiority; p = 0.921, t-test, 2 sided
Statistical Analysis 17: Comparison: Chronic Kidney Disease vs Age Matched Control; This compares the 12 month CRPWV measure of the CKD and Control groups; Test type: Superiority; p = 0.887, t-test, 2 sided
Statistical Analysis 18: Comparison: Chronic Kidney Disease vs Age Matched Control; This compares the 12 month CFPWV measure of the CKD and Control groups; Test type: Superiority; p = 0.759, t-test, 2 sided
Statistical Analysis 19: Comparison: Age Matched Control; This compares the baseline and 12 month CBPWV measure of the Control groups; Test type: Superiority; p = 0.851, t-test, 2 sided
Statistical Analysis 20: Comparison: Age Matched Control; This compares the baseline and 12 month CRPWV measure of the Control groups; Test type: Superiority; p = 0.733, t-test, 2 sided
Statistical Analysis 21: Comparison: Age Matched Control; This compares the baseline and 12 month CFPWV measure of the Control groups; Test type: Superiority; p = 0.902, t-test, 2 sided
Statistical Analysis 22: Comparison: Chronic Kidney Disease-ACE-I vs Chronic Kidney Disease; This compares the 12 month CBPWV measure between the CKD ACE-I and CKD Control groups; Test type: Superiority; p = 0.414, t-test, 2 sided
Statistical Analysis 23: Comparison: Chronic Kidney Disease-ACE-I vs Chronic Kidney Disease; This compares the 12 month CRPWV measure between the CKD ACE-I and CKD Control groups; Test type: Superiority; p = 0.942, t-test, 2 sided
Statistical Analysis 24: Comparison: Chronic Kidney Disease-ACE-I vs Chronic Kidney Disease; This compares the 12 month CFPWV measure between the CKD ACE-I and CKD Control groups; Test type: Superiority; p = 0.990, t-test, 2 sided
Statistical Analysis 25: Comparison: Age Matched Control-ACE-I vs Age Matched Control; This compares the 12 month CBPWV measure between the ACE-I Control and CKD Control groups; Test type: Superiority; p = 0.273, t-test, 2 sided
Statistical Analysis 26: Comparison: Age Matched Control-ACE-I vs Age Matched Control; This compares the 12 month CRPWV measure between the ACE-I Control and CKD Control groups; Test type: Superiority; p = 0.516, t-test, 2 sided
Statistical Analysis 27: Comparison: Age Matched Control-ACE-I vs Age Matched Control; This compares the 12 month CFPWV measure between the ACE-I Control and CKD Control groups; Test type: Superiority; p = 0.102, t-test, 2 sided

3. Secondary Outcome: Change in Blood Pressure From Baseline to 12 Months
Description: Change in Blood Pressure will be used to measure the effect of ACE-inhibitors on the clinical markers of Cardiovascular Disease in participants with stage 3 CKD.
Time Frame: up to 12 months
Population: There is limited data for this study, the PI is now in private practice and the raw data no longer exists to answer this outcome. We have done our due diligence to populate this record with data that remains.
Arm/Group | Chronic Kidney Disease-ACE-I | Chronic Kidney Disease | Age Matched Control-ACE-I | Age Matched Control
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 12 months
Description: There is limited data for this study, the PI is now in private practice and unreachable. The remaining study team has found data only in support of Aim 1 (CKD aortic stiffness vs healthy controls), no data for ACE-I arms.
Arm/Group | Chronic Kidney Disease-ACE-I | Chronic Kidney Disease | Age Matched Control-ACE-I | Age Matched Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/17 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/17 | 0/14
Other Adverse Events (participants affected / at risk) | 2/8 | 1/4 | 3/17 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease-ACE-I (N=8) | Chronic Kidney Disease (N=4) | Age Matched Control-ACE-I (N=17) | Age Matched Control (N=14)
Uticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Lip Parasthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Headache (General disorders) | 0 | 0 | 1 | 0
Stiff Neck (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Low Blood Pressure (Vascular disorders) | 0 | 0 | 1 | 0
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
There is limited data for this study, the PI is now in private practice and some raw data no longer exists to answer this outcome. We have done our due diligence to populate this record with data that remains.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes